CLINICAL TRIAL: NCT01726790
Title: Effect of Intravitreal Bevacizumab on Corneal Endothelium
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Kasem Yospaiboon, Kasem Yospaiboon, MD, Khon Kaen University
Other Study IDs: HE541020
Record Dates: First submitted 2012-11-11; First posted 2012-11-15 (Estimated); Last update posted 2012-11-15 (Estimated); Status verified 2012-11

CONDITIONS: Corneal Endothelial Cell Loss
Keywords: corneal endothelium; Bevacizumab; Intravitreal injection; Confoscan
MeSH Terms: conditions — Corneal Endothelial Cell Loss

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To evaluate corneal endothelium cell change after intravitreal Bevacizumab injection

DETAILED DESCRIPTION:
Intravitreal Bevacizumab has been used by retinal specialist in treatment many retinal diseases. Although it not approved by FDA for treatment. In many In vitro studies, its showed saftey in the eyes especially for corneal endothelium cells, that important cells to keep cornea clear. This study use Confoscan-Corneal confocal microsope to evaluate corneal endothelium before and after intravitreal Bevacizumab injection in routine retinal disease at 6 month follow up.

ELIGIBILITY:
Inclusion Criteria:

* aged between 20 and 80 years old
* can come to regular follow up at 6 month
* signed written consent forms
* not have corneal scar, or glaucoma
* history of treatment with laser or anti-VEGF therapy in 3 month prior to recruit
* high risk in cerebrovascular and cardiovascular diseases
* Pregnancy and breastfeeding
* can undergo confocal microspopy

Exclusion Criteria:

* History of intraocular surgery or ocular trauma during study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient in retinalvascular clinic with diagnosis of retinal vein occlusion with macular edema, diabetic macular edema, wet aged related macular degeneration and submacular hemorrhage)treated with intravitreal Bevacizumab
Sampling Method: Non-Probability Sample
Enrollment: 37 (Estimated)
Dates: Start 2011-08; Primary Completion 2013-06 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Corneal endothelium cell change after intravitreal Bevacizumab injection | 6 months
  Measure the corneal endothelium cell using Confoscan4-Corneal confocal microscope in patient in retinal vascular clinic before and after treat with intravitreal Bevacizumab

SECONDARY OUTCOMES:
Assess the complication after intravitreal Bevacizumab injection | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- KKU eye center, department of Ophthalmolgy, faculty of medicine, khon kaen university, Khon Kaen, Changwat Khon Kaen, Thailand